CLINICAL TRIAL: NCT02580045
Title: CSF Pharmacokinetics of Systemic Anti-Cancer Therapies in Patients With Advanced Cancer
Brief Title: Pharmacokinetics of Systemic Anti-Cancer Therapies in the Cerebrospinal Fluid (CSF) of Patients With Advanced Cancer
Status: Terminated | Type: Observational
Why Stopped: Inadequate Accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00062142
Record Dates: First submitted 2015-10-07; First posted 2015-10-20 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Cancer Patients on an Anti-cancer Therapy; Advanced Cancer; Brain Metastasis
Keywords: metastatic cancer; lumbar puncture; advanced cancer; brain metastases; chemotherapy; endocrine therapy; HER2 targeted therapy; immune therapy; anti-cancer therapy; blood brain barrier; pharmacokinetics; Duke University; brain metastasis
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples and cerebrospinal fluid samples are to be collected for pharmacokinetic analysis by blood draw and lumbar puncture, respectively.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This clinical trial is being done to learn more about how different types of cancer treatments affect cancer cells when they spread to the brain. Many cancer treatments are not able to make their way into the brain or into spinal fluid of the central nervous system. This is because they cannot cross what is called the "blood-brain barrier" or "BBB". The BBB is like a protective shield that only allows certain materials pass through to reach the brain but not others. This study is being initiated to help researchers learn more about what types of cancer treatments make it through the BBB to attack cancer cells within the brain, and what treatments do not make it through the BBB. Learning more about this may help future researchers develop more effective cancer drugs that better fight cancer cells that have spread to the brain.

DETAILED DESCRIPTION:
Very little is known about the penetration of systemic therapies through the normal blood brain barrier and the ways in which a brain metastasis or radiation would impact the permeability of the blood brain barrier. This study would be one of the first to examine the concentrations of systemic cancer therapies in the cerebrospinal fluid (CSF) with matched serum samples. Additionally, the concentration of these therapies in brain metastasis surgical specimens would be of particular interest to correlate with serum and CSF levels, length of time on therapy, and latency to developing brain metastases in future studies.

As participants in this study, patients scheduled for a lumbar puncture per their standard of care treatment will be subject to a withdrawal of 15cc's of cerebrospinal fluid for pharmacokinetic analysis. They will also have a blood draw of 5mL within 2 hours of the lumbar puncture for serum pharmacokinetics. If the patient is eligible for and elects to proceed with surgical resection of a brain metastasis, optional CSF and serum samples would be drawn at the time of resection.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic cancer patients on systemic anti-cancer therapy (chemotherapy, endocrine therapy, HER2 targeted therapy, immune therapy).
2. Patients must be able to have a lumbar puncture within 2 half-lives of the last dose of systemic therapy.
3. Patients undergoing an LP for any reason with known advanced cancer on systemic anti-cancer therapy are eligible.
4. Patients with new or previously treated brain metastases are eligible.
5. Patients may have received prior stereotactic radiosurgery to the brain and/or whole brain radiation.
6. No limitations on prior systemic or intrathecal therapies.
7. There are no restrictions on systemic therapy at enrollment.
8. Laboratory criteria: normal renal function: creatinine < 1.5 x upper limit of normal (ULN)), liver function: bilirubin < 1.5 x ULN, transaminases < 2 x ULN, except in known hepatic disease, wherein may be < 5 x ULN, and blood counts: WBC ≥ 2.0, Neutrophils ≥1500, platelets ≥100,000, Hemoglobin ≥ 10.
9. Age > 18 years
10. Patients must have the ability to give informed consent.
11. Patients must have a signed informed consent form prior to enrollment on study.

Exclusion Criteria:

1. No history of lumbar surgery or other pre-existing spinal conditions that would preclude a safe, reliable lumbar puncture.
2. Patients should have no significant psychiatric illness or medical illness that would preclude the ability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic or advanced cancer patients on systemic anti-cancer therapy including chemotherapy, endocrine therapy, HER2-targeted therapy, and immune therapy.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
The concentration of drug metabolites of systemic anti-cancer therapies in the cerebrospinal fluid | up to 3 weeks
  CSF pharmacokinetics of systemic anti-cancer therapies, as measured by the concentration of their metabolites in the cerebrospinal fluid, will be obtained via lumbar puncture. The lumbar puncture will take place within 2 half-lives of the last dose of systemic therapy. Because a wide variety of anti-cancer therapies will be studied in this trial, there is significant variability in the half-lives of these therapies. Some will take place 2-24 hours after the last dose of systemic therapy. Some will take place 1-6 days after the last dose of systemic therapy. Some will take place 1-3 weeks after the last dose of systemic therapy. The time of the lumbar puncture procedure will depend greatly on the identity of the systemic therapy with which the subject is being treated. In patients undergoing surgical resection of a brain metastasis, an additional CSF sample is optional.
Ratio of serum to CSF concentration of systemic anti-cancer therapies as measured by concentration of drug metabolites in serum and in CSF | up to 3 weeks
  CSF and serum pharmacokinetics of systemic anti-cancer therapies, as measured by the concentration of their metabolites, will be obtained via lumbar puncture and blood draw, respectively. The lumbar puncture and blood draw will take place together within 2 half-lives of the last dose of systemic therapy. Because a wide variety of anti-cancer therapies will be studied in this trial, there is significant variability in the half-lives of these therapies. Some will take place 2-24 hours after the last dose of systemic therapy. Some will take place 1-6 days after the last dose. Some will take place 1-3 weeks after the last dose. The time of the lumbar puncture procedure will depend greatly on the identity of the systemic therapy with which the subject is being treated. In patients undergoing surgical resection of a brain metastasis, an additional matched CSF and serum sample is optional.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly L Blackwell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States